CLINICAL TRIAL: NCT03196960
Title: Effects of Mobility Dose in Surgical Intensive Care Unit Patients on Adverse Discharge Disposition
Brief Title: Effects of Mobility Dose in Surgical Intensive Care Unit Patients
Acronym: MQS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Technical University of Munich (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, MD PhD, Associate Professor of Anaesthesia, Harvard Medical School; Clinical Director, Critical Care Division, Massachusetts General Hospital
Other Study IDs: 2016P002045
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Sarcopenia; Muscle Weakness; Critical Illness
Keywords: Mobilization Therapy; Critical Illness; Muscle Strength; Functional Mobility; Outcome; Intensive Care Unit; Quality of Life
MeSH Terms: conditions — Sarcopenia; Muscle Weakness; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to assess if the mobility dose that patients receive in the surgical intensive care unit (SICU) predicts adverse discharge disposition (primary endpoint), and muscle wasting diagnosed by bedside ultrasound (secondary endpoint).

DETAILED DESCRIPTION:
Our research group aims to better understand how patients on the SICU are mobilized and the impact it has on adverse discharge disposition and functional outcome after hospital discharge.

We have previously developed and validated the Surgical Intensive Care Unit Optimal Mobilization Score (SOMS), an algorithm to guide and facilitate early mobilization to advance mobility of SICU patients (NCT01363102). In addition, we have established the use of bedside ultrasound technology to quantify cross sectional area of the rectus femoris muscle, which allows an objective, user-independent quantification of muscle wasting (NCT02270502).

In this study we measure the dose of mobility, defined as a function of both the mobility provided by nursing and physical therapists (e.g., sitting at the edge of the bed, ambulating) as well as its duration. We will build on an existing mobility intensity quantification tool (NCT01674608) and add a domain that quantifies its duration in order to obtain a broad picture of the mobilization of patients on the SICU. The mobility dose is expressed by the mobility quantification score that has been developed by our team. We will then test the hypotheses that mobilization dose in the ICU predicts discharge disposition, defined as discharge to facilities providing long-term care assistance for daily activities, including nursing homes and skilled nursing facilities, hospice at the patient's home, hospice in a health care facility; or in-hospital mortality. Further we will evaluate the association between mobility dose and cross sectional area of the rectus femoris muscle measured by bedside ultrasound as a potential reflection of ICU-acquired muscle weakness (exploratory outcome).

Mobilization Quantification score: MQS (Detailed table linked in reference section)

This score integrates the highest rated activities within each mobility session - from physical therapy and nursing. By multiplying the scale it gets greater and allows a better interpretation of mobility intensity. It adds value of mobility dose across sessions considering the entire spectrum of active participation of the patient over the day.

Some specifics:

* If patient achieves a level in between predefined MQS levels we score the closest lower level
* We collect mobility data for the night time by interviewing the day nurses and asking them about the patients' mobilization also during night time
* We round up the duration of each mobility session: Passive range of motion (PRM) conducted 4 times during the day counts as: 1*4=4 (corresponding to 4 units/hours)
* For each session, we calculate the highest mobility level for the duration of the mobility session: e.g. Patient is standing for 5 minutes before s/he walks with 2 assists for 10 minutes: 3*7=21 (adding up the duration of various activities within a session and multiplying it by the highest achieved mobility level). Sitting passively in the chair is an exception (see below).

Sitting:

* Sitting in the chair counts as a separate session. Per sitting session a maximum of 2 hours are counted. For example: if a patient was sitting for a duration of either 2, 4 or 5 hours, we would always count: 2*4=8
* For patients stepping/shuffling/walking to the chair we use level 5 every time the patient is doing it. E.g. patient is shuffling to the chair, sitting for 2 hours and then walking back: 5*1+2*4+5*1 =28
* Distinct sitting sessions are defined by the patient being back in bed in between the sessions of sitting in the chair. E.g. the patient gets actively to chair by stand-step/shuffle, sits in chair for 6 hours, during sitting session patient gets up twice and afterwards gets back to bed by stand-step/shuffle:

5*1(to chair)+2*4(sitting)+5*1(back to bed)+5*2(standing up 2x in between)=28

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or greater)
* Barthel score ≥70 from a proxy describing patient function 2 weeks before admission
* Expected stay on the ICU of >=3 days

Exclusion Criteria:

* Patients transferred from other hospitals, long-term rehabilitation facilities or nursing homes with a preceding stay of more than 48 hours
* Hospitalization 1 month prior to ICU admission >7 days
* Discussion about changing the goals of care from cure to comfort
* High risk of persistent brain injury (GCS<5 motor component and presence of TBI)
* Patients with neurodegenerative diseases
* Subjects with absence of a lower extremity
* Patients with paraplegia or tetraplegia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients recovering in an intensive care unit following a trauma or a surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Hospital Discharge Disposition | Patient will be followed until hospital discharge, an expected 3 to 30 days
  Adverse hospital discharge is defined as discharge to facilities providing long-term care assistance for daily activities, including nursing homes and skilled nursing facilities, hospice at the patient's home, hospice in a health care facility, or in-hospital mortality.

SECONDARY OUTCOMES:
Rectus Femoris Muscle Cross Sectional Area | Rectus femoris cross sectional area will be measured twice, at enrollment and day of ICU discharge, an expected 3 to 30 days.
  Rectus femoris cross sectional area will be measured by bedside ultrasound
Mobility Dose as measured by the Mobilization Quantification Score (MQS) | Patients will be followed until SICU discharge, an expected 3 to 30 days.
  Mobilization Quantification Score (MQS) is a composition of the validated ICU mobility score, a 0 to 10 value scale that measures the mobility milestones in critically ill patients, multiplied by a for each level previously defined time unit (5 or 30 minutes correspond to one unit).
Abbreviated Functional independence measure (FIM) score at Surgical Intensive Care Unit (SICU) discharge and hospital discharge | Patients will be followed until hospital discharge an expected 3 to 40 days.
  Abbreviated FIM score obtained by physical therapy (PT) within 48 hours of discharge, and by research assistant on the day of discharge if the subject was not seen by PT in the indicated time period.
SICU length of stay | Patients will be followed until SICU discharge, an expected 3 to 30 days.
  Number of days from SICU admission to SICU discharge
Hospital length of stay | Patients will be followed until hospital discharge an expected 3 to 40 days.
  Number of days from hospital admission to hospital discharge
SICU Ventilator-free days | Patients will be followed until ICU discharge, an expected 3 to 30 days.
  Number of days spent on the SICU that patient is not receiving mechanical ventilation.
SICU Vasopressor-free days | Patients will be followed until ICU discharge, an expected 3 to 30 days.
  Number of days spent on the SICU that patient is not receiving any vasopressor medications.
SICU Delirium-free days | Patients will be followed until ICU discharge, an expected 3 to 30 days.
  Days spent on the SICU that patient is Confusion assessment method (CAM)-ICU/Richmond Agitation-Sedation Scale (RASS) negative.
SICU Neuromuscular Blocking drug-free days | Patients will be followed until ICU discharge, an expected 3 to 30 days.
  Number of days spent on the ICU that patient is not receiving Neuromuscular Blocking Agents
Opioid Use | Patients will be followed until ICU discharge, an expected 3 to 30 days.
  Opioid dose administered, calculated as morphine equivalent dose.
Corticosteroid Days | Patients will be followed until ICU discharge, an expected 3 to 30 days.
  Number of day on ICU with corticosteroid administration Number of day on ICU with corticosteroid administration Number of ICU days with corticosteroid administration
Physical Work Capacity | Measured three months after hospital discharge
  Obtained after hospital discharge, measured by the Duke Activity Status Index (DASI)
3-Month Mortality | Evaluated three months after hospital discharge
Falls | Patients will be followed until ICU discharge, an expected 3 to 30 days.
  Number of Falls during ICU stay
Side effects of mobilization therapy | Patients will be followed until ICU discharge, an expected 3 to 30 days.
  Number of unfavorable signs and symptoms or unintended deterioration of clinical status associated with mobilization therapy, including, but not limited to, unplanned extubation or dislodgment of drains, arterial catheters, venous devices, or other medical equipment. The relationship of any untoward event to mobilization therapy was assessed by the clinician and reported as unrelated, unlikely, possibly, or definitely related. Adverse events (AE) were also categorized by intensity as mild, moderate, or severe

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Klinikum Rechts der Isar, Munich, Bavaria, Germany
- Università degli Studi di Brescia, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mueller N, Murthy S, Tainter CR, Lee J, Riddell K, Fintelmann FJ, Grabitz SD, Timm FP, Levi B, Kurth T, Eikermann M. Can Sarcopenia Quantified by Ultrasound of the Rectus Femoris Muscle Predict Adverse Outcome of Surgical Intensive Care Unit Patients as well as Frailty? A Prospective, Observational Cohort Study. Ann Surg. 2016 Dec;264(6):1116-1124. doi: 10.1097/SLA.0000000000001546. PMID 26655919
- [Background] Schaller SJ, Anstey M, Blobner M, Edrich T, Grabitz SD, Gradwohl-Matis I, Heim M, Houle T, Kurth T, Latronico N, Lee J, Meyer MJ, Peponis T, Talmor D, Velmahos GC, Waak K, Walz JM, Zafonte R, Eikermann M; International Early SOMS-guided Mobilization Research Initiative. Early, goal-directed mobilisation in the surgical intensive care unit: a randomised controlled trial. Lancet. 2016 Oct 1;388(10052):1377-1388. doi: 10.1016/S0140-6736(16)31637-3. PMID 27707496
- [Background] Lee JJ, Waak K, Grosse-Sundrup M, Xue F, Lee J, Chipman D, Ryan C, Bittner EA, Schmidt U, Eikermann M. Global muscle strength but not grip strength predicts mortality and length of stay in a general population in a surgical intensive care unit. Phys Ther. 2012 Dec;92(12):1546-55. doi: 10.2522/ptj.20110403. Epub 2012 Sep 13. PMID 22976446
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Kasotakis G, Schmidt U, Perry D, Grosse-Sundrup M, Benjamin J, Ryan C, Tully S, Hirschberg R, Waak K, Velmahos G, Bittner EA, Zafonte R, Cobb JP, Eikermann M. The surgical intensive care unit optimal mobility score predicts mortality and length of stay. Crit Care Med. 2012 Apr;40(4):1122-8. doi: 10.1097/CCM.0b013e3182376e6d. PMID 22067629
- [Background] Tipping CJ, Bailey MJ, Bellomo R, Berney S, Buhr H, Denehy L, Harrold M, Holland A, Higgins AM, Iwashyna TJ, Needham D, Presneill J, Saxena M, Skinner EH, Webb S, Young P, Zanni J, Hodgson CL. The ICU Mobility Scale Has Construct and Predictive Validity and Is Responsive. A Multicenter Observational Study. Ann Am Thorac Soc. 2016 Jun;13(6):887-93. doi: 10.1513/AnnalsATS.201510-717OC. PMID 27015233
- [Derived] Scheffenbichler FT, Teja B, Wongtangman K, Mazwi N, Waak K, Schaller SJ, Xu X, Barbieri S, Fagoni N, Cassavaugh J, Blobner M, Hodgson CL, Latronico N, Eikermann M. Effects of the Level and Duration of Mobilization Therapy in the Surgical ICU on the Loss of the Ability to Live Independently: An International Prospective Cohort Study. Crit Care Med. 2021 Mar 1;49(3):e247-e257. doi: 10.1097/CCM.0000000000004808. PMID 33416257
- Available data/document: Scoring Sheet — https://docs.google.com/document/d/1pqYbMe4S-W-vgYRHzd1d4Is7s6ZbMt_MGDlWtndRRdM/edit?usp=sharing — Mobilization Quantification Score

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03196960/SAP_000.pdf